CLINICAL TRIAL: NCT06620250
Title: A Randomized Controlled Trial：a Study of the Impact of Digital Intervention on Parents/primary Caregivers' Myopia Prevention and Control Health Literacy on Preschoolers' Myopia and Physical and Mental Health
Brief Title: A Study of the Impact of Digital Intervention on Parents/primary Caregivers' Myopia Prevention and Control Health Literacy on Preschoolers' Myopia and Physical and Mental Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20240808
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Myopia; Mental Health; Obesity
MeSH Terms: conditions — Myopia; Psychological Well-Being; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Prevention and control of myopia (Experimental): two articles per month were sent to the parent/primary caregiver for acceptance of the intervention, and one month after the intervention began, an"Expert said" video intervention was added, at the beginning of each month, a video was posted for them to learn; three months after the start of the intervention, the wechat message intervention was added, and relevant knowledge about myopia prevention and control was sent to the wechat group every Tuesday morning; nine months after the start of the intervention, increase the text message intervention, send text messages every Friday evening to remind children of the weekend outdoor activities. In addition, live broadcasts will be held in March September and June 6 to answer parents' questions and concerns.
  Interventions: Combination Product: Digital Prevention and control of myopia
- Control Group (No Intervention): No intervention of any kind

INTERVENTIONS:
Combination Product: Digital Prevention and control of myopia — The Digital Intervention Programme for parents/primary caregivers is primarily a digital intervention to address the attitudes, knowledge and actions of parents or primary caregivers of pre-school children regarding the prevention and control of myopia.
  Arms: Digital Prevention and control of myopia

SUMMARY:
The study is a Randomized controlled trial based on digital interventions, involving pre-school children and their parents or major caregivers. To compare the myopia and physical and mental health status of preschool children before and after intervention between intervention group and control group, to confirm the effect of digital intervention on prevention and control of Myopia and physical and mental health of preschool children.

DETAILED DESCRIPTION:
In this study, wechat, online courses, live broadcast and SMS were used to transfer the knowledge of myopia prevention and control to parents/primary caregivers, and to promote their attitude and behavior change. The intervention period was from October to December 2025. The control group did not 2024 any intervention. The prevention and control of Myopia and health literacy of the parents and main adopters were collected at baseline and after the intervention respectively, visual data and physical and mental health status of preschool children were collected every six months.

ELIGIBILITY:
Inclusion Criteria:

* No cognitive impairment and communication impairment
* Volunteer and sign the informed consent
* Fill in the questionnaire
* Skilled in using electronic equipment

Exclusion Criteria:

* Children with congenital glaucoma, cataract, strabismus and other congenital eye diseases
* Children with a history of ocular trauma, eye surgery, or complications of myopia
* Do not cooperate with the investigation

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 882 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevention and control of Myopia Health Literacy Rating Scale | 0,6month，12month
  The scale was used to assess the prevention and control of myopia health literacy of parents/primary caregivers, including 3 dimensions, 6 aspects and 31 items, each with 3 or 5 options. The forward score was 1,2,3,4,5(1,2,3) , and the reverse score was 5,4,3,2,1(3,2,1) . The scale scores ranged from 0 to 102, the higher the score, the higher the health literacy of prevention and control of myopia.
Myopia screening | 0,6month,12month
  Myopia screening includes Naked Eye Far Vision Examination, computer optometry and axial length measurement.In the state of non-ciliary paralysis, SE ≤ -0.50 D, visual acuity ≤4.7 at 3 years old, 4.8 at 4 years old, 4.9 at 5 years old, and less than 5.0 in the naked eye of children and adolescents over 6 years old were considered as screening myopia.
BMI | 0, 6month，12month
  BMI = weight (kg)/[ height (m)]2. The standard deviation method was used to evaluate the physical growth of children（WS/T 423-2022）, + 1 SD≤ age BMI ≤ + 2 SD was defined as overweight, + 2 SD ≤ age BMI≤ + 3 SD was defined as Obesity.
Strength and Difficulties Questionnaire | 0,6month,12month
  The mental health status of preschool children was evaluated by Strength and Difficulties Questionnaire, SDQ，SDQ includes 5 dimensions: emotional symptoms, conduct problems, hyperactivity problems, peer interaction problems and prosocial behaviors.The questionnaire was scored on a 3-point scale, and was evaluated from non-conformity (0 points) to full conformity (2 points) . The scale scores ranged from 0 to 40, the higher the score, the more serious the emotional and behavioral problems.